CLINICAL TRIAL: NCT05565937
Title: A Safety and Effectiveness Study of a Contact Lens Cleaning and Disinfecting Solution
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Contact Lens Cleaning and Disinfecting Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 914
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Refractive Ametropia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BL-3100-NBR03 (Experimental): BL-3100-NBR03 multi-purpose solution
  Interventions: Device: BL-3100-NBR03 multi-purpose solution
- renu® Advanced Formula (Active Comparator): renu® Advanced Formula multi-purpose solution
  Interventions: Device: renu® Advanced Formula multi-purpose solution

INTERVENTIONS:
Device: BL-3100-NBR03 multi-purpose solution — BL-3100-NBR03 multi-purpose solution used to clean and disinfect contact lenses
  Arms: BL-3100-NBR03
Device: renu® Advanced Formula multi-purpose solution — renu® Advanced Formula multi-purpose solution used to clean and disinfect contact lenses
  Arms: renu® Advanced Formula

SUMMARY:
Approximately 340 participants (680 eyes) will be enrolled in this three-month, two-arm, 1:1 randomized, parallel-group, bilateral, double-masked study at approximately 22 investigative sites in the United States. Participants will be required to wear dispensed study lenses on a daily wear basis for three months with scheduled in-office replacement of study lenses at the 1-Month and 2-Month Follow-Up Visits.

ELIGIBILITY:
Inclusion Criteria:

1. Is of legal age (at least 18) on the date the Informed Consent Form (ICF) is signed
2. Is able to read, understand, and provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide authorization as appropriate for local privacy regulations
3. Is a habitual wearer (at least 3 months)
4. Has typically cleaned and disinfected their pre-study contact lenses daily
5. Must have spectacle correctable distance visual acuity through spherocylindrical refraction to 40 letters (0.14 logarithm of the minimal angle of resolution (logMAR) or better in each eye, at 2 meters distance with high contrast chart
6. Has clear central corneas and is free of any anterior segment disorders
7. Is a habitual user of a lens care product for cleaning, disinfecting, and storage of lenses
8. Requires lens correction in both eyes
9. Wears the same manufacturer and brand of lens in both eyes
10. Agrees to wear study lenses on a daily wear basis for approximately three months
11. Is willing and able to comply with all treatment and follow-up/study procedures.

Exclusion Criteria:

1. Is currently using a hydrogen-peroxide cleaning and disinfecting solution
2. Participated in any drug or device clinical investigation within 30 days prior to entry into this study
3. Is a female of childbearing potential (those who are not surgically sterilized or postmenopausal) if they meet any one of the following conditions:

   * they are currently pregnant
   * they plan to become pregnant during the study
   * they are breastfeeding
4. Has worn gas permeable (GP) lenses within the last 30 days
5. Has worn polymethylmethacrylate (PMMA) lenses within the last three months
6. Has typically worn their pre-study contact lenses on an extended wear basis, sleeping in their lenses one night or more per week, during the last year
7. Has any systemic disease currently affecting ocular health or which in the Investigator's opinion may have an effect on ocular health during the course of the study
8. Subjects with an active ocular disease, or who are using any ocular medication.
9. Is using any medications that will, in the Investigator's opinion, affect ocular physiology or lens performance
10. Currently wears monovision, multifocal, or toric contact lenses
11. Has ocular astigmatism of 1.00D or greater in either eye
12. Has anisometropia (spherical equivalent) of greater than 2.00D
13. Has any grade 2 or greater finding during the slit-lamp examination (refer to Appendix B for Methods of Clinical Evaluation)
14. Has corneal infiltrates, of ANY GRADE
15. Has any "Present" ungraded finding during the slit-lamp examination (refer to Appendix B for Methods of Clinical Evaluation) that, in the Investigator's judgment, interferes with contact lens wear.
16. Has typically worn their pr-study control lenses on an extended wear bases, sleeping on their lenses one night or more per week, during the last year.
17. Is aphakic
18. Is amblyopic
19. Has had any corneal surgery (e.g., refractive surgery)
20. Is allergic to any component in the study care products.
21. Is an employee of any of the study investigative sites or a family member of an employee of the investigative site, including family members living outside of the employee's household
22. Is an Ophthalmologist, an Optometrist, an Optician, or an Ophthalmic Assistant/Technician, or currently resides with a person with any of these specialties
23. Is an employee of a manufacturer of contact lenses or contact lens care products (e.g., Alcon, Bausch + Lomb, Ciba Vision, CooperVision, Vistakon, Johnson & Johnson, etc.) or currently resides with a person employed by any of these manufacturers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Donatello, Study Director — Bausch & Lomb Incorporated
Locations (19):
- United States (19):
  - Eric White OD Inc, San Diego, California
  - Lee & Woo Optometry, San Francisco, California
  - Chester T Roe III MD Prof LLC, Denver, Colorado
  - Eola Eyes, Orlando, Florida
  - Golden Vision, Sarasota, Florida
  - The Eyecare Studio, LLC, Decatur, Georgia
  - Kannarr EyeCare, Pittsburg, Kansas
  - Casco Bay EyeCare, Portland, Maine
  - Complete Eye Care of Medina, Medina, Minnesota
  - Advanced Eye Care, PC, Raytown, Missouri
  - Koetting Associates, St Louis, Missouri
  - InSight Eyecare, Warrensburg, Missouri
  - Berlin Eyecare Associates, West Berlin, New Jersey
  - Spectrum Eyecare, Jamestown, New York
  - Saccco Eye Group, Vestal, New York
  - Oculus Research, Raleigh, North Carolina
  - Total Eye Care, PA, Memphis, Tennessee
  - Optometric Physicians of Middle Tennessee, Nashville, Tennessee
  - Biopharma Informatic, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
Started | 143 | 152 (1 subject in the renu advance formula was not dispensed study product and is not included in the safety analysis)
Completed | 140 | 147
Not Completed | 3 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Persistent study-related symptoms /complaints | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Pregnancy | 0 | 2
Not completed — Anisometropia | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula | Total
Number analyzed (Participants) | 143 | 152 | 295
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (10.26) | 37.5 (9.84) | 36.5 (10.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 109 | 209
  Male | 43 | 43 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 134 | 146 | 280
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 17 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 13 | 16 | 29
  White | 109 | 112 | 221
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 143 | 152 | 295

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Averaged Over All Follow-up Visits
Description: Overall comfort will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response
Time Frame: Assessed at all follow-up visits through 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
Number analyzed (Participants) | 143 | 152
Number analyzed (Eyes) | 286 | 304
score on a scale | 91.7 (9.99) | 90.7 (10.83)

2. Primary Outcome: Vision Averaged Over All Follow-up Visits
Description: Vision will be assessed for each eye on a scale from 0 to 100, with 100 denoting the most favorable response
Time Frame: Assessed at all follow-up visits through 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
Number analyzed (Participants) | 143 | 152
Number analyzed (Eyes) | 286 | 304
score on a scale | 95.5 (6.69) | 94.3 (7.75)

3. Primary Outcome: The Proportion of Eyes With a Maximum Degree of Front Surface Deposits Grade of <= 2 Over All Follow-up Visits With 0 Being Absent of Deposits.
Description: The degree of front surface deposits will be graded for each eye as:
  0 - Absent, clean surface.
  1. - Very slight, only visible after tear film drying.
  2. - Slight, visible deposits easily removable.
  3. - Moderate, deposits adherent and not removable.
  4. - Severe, non-removable deposits and comfort affected.
Time Frame: Assessed at all follow-up visits through 3 months.
Population: All randomized subjects with at least one non-missing values for front surface deposit grading. Two subjects (4 eyes) in the BL-3100-NBR03 arm and 1 subject (2 eyes) in the renu Advanced Formula arm with no front surface grading measurements reported were excluded from this analysis.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
Number analyzed (Participants) | 141 | 151
Number analyzed (Eyes) | 282 | 302
percentage of eyes
  The Percentage of Eyes with Front Surface Deposits Grade of <= 2 | 99.3 | 97.7
  The Percentage of Eyes with Front Surface Deposits Grade of >2 | 0.7 | 2.3

4. Primary Outcome: The Proportion of Eyes With Any Slit-lamp Findings Greater Than Grade 2 Over All Follow-up Visits.
Description: Graded slit-lamp findings will be assessed for each eye using Grades 0 through 4.
Time Frame: Assessed at 3 months
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
Number analyzed (Participants) | 143 | 151
Number analyzed (Eyes) | 282 | 302
percentage of eyes
  Present | 0 | 0.7
  Absent | 100 | 99.3

ADVERSE EVENTS:
Time Frame: AE data collected over all scheduled follow-up visits approximately 3 months
Arm/Group | BL-3100-NBR03 | Renu® Advanced Formula
All-Cause Mortality (participants affected / at risk) | 0/143 | 0/151
Serious Adverse Events (participants affected / at risk) | 0/143 | 1/151
Other Adverse Events (participants affected / at risk) | 0/143 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BL-3100-NBR03 (N=143) | Renu® Advanced Formula (N=151)
Appendicitis (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT05565937/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT05565937/SAP_001.pdf